CLINICAL TRIAL: NCT00358527
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Multicenter Study of Mometasone Furoate Nasal Spray on Sleep Disturbances and Daytime Somnolence in Subjects With Symptomatic Seasonal Allergic Rhinitis
Brief Title: Mometasone Furoate on Sleep Disturbances in Subjects With Seasonal Allergic Rhinitis (Study P04608) (COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04608
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate Nasal Spray (Experimental): Mometasone Furoate Nasal Spray 200 mcg, once daily.
  Interventions: Drug: Mometasone Furoate Nasal Spray (MFNS)
- Matching placebo nasal spray (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray (MFNS) — MFNS 50 mcg/spray: self-administered, two sprays per nostril (ie, 200 mcg QD), once daily (each morning), for 28 days.
  Other Names: MFNS
  Arms: Mometasone Furoate Nasal Spray
Other: Placebo — Matching placebo nasal spray: 2 sprays per nostril once daily for 28 days
  Arms: Matching placebo nasal spray

SUMMARY:
This study will hope to show that by relieving the participant's nasal symptoms of seasonal allergies using mometasone furoate nasal spray, the participant will obtain a better quality of night-time sleep, which in turn, causes less daytime sleepiness so that he/she can function productively during the day.

ELIGIBILITY:
Inclusion Criteria:

* Must be >=18 years of age and older, of either sex, and of any race.
* Clinically symptomatic at Screening (Day -7 to -4)and at Baseline (Day 1)
* At Screening Visit, must have complaints of sleep disturbance while symptomatic with seasonal allergic rhinitis (SAR) and must have a score of 30 or greater for the Sleep Disturbance Sleep Scale (items 1,3,7 and 8)
* At the Baseline Visit, must have complaints of sleep disturbance and daytime somnolence while symptomatic with SAR and with a score of 30 or greater for the Sleep Problems Index II (SLP9) and 30 or greater for the Daytime Somnolence Sleep Scale (items 6, 9, and 11)
* Must have a 2-year or longer history of SAR occurring during the same season as the current study.
* Must have skin tests positive for outdoor allergens common in subjects with SAR prevalent during the time of this study, such as, trees, grasses, weeds, ragweed, and molds. The skin tests should be performed at Screening if not done within 12 months prior to the Screening Visit
* Must be free of clinically significant disease that would interfere with study evaluations
* Women of childbearing potential need to use a medically accepted method of birth control prior to Screening and during the study, or provide documentation of surgical sterilization. Women who are not sexually active at enrollment must consent to the use of a medically accepted method of birth control if/when they become sexually active during study participation.
* Female subjects of childbearing potential must have a negative urine pregnancy test at the time of enrollment at the Baseline Visit.

Exclusion Criteria:

* Women who are pregnant, intend to become pregnant during the study, or are nursing
* Evidence of nasal polyps, deviated septum, or other intranasal anatomical obstruction(s) that would interfere with nasal airflow
* Acute or chronic sinusitis being treated with antibiotics and/or topical or oral nasal decongestants
* Acute respiratory infection within 2 weeks of the Screening Visit
* Diagnosis of clinically relevant sleep problems unassociated with allergies
* Complaints (within 12 months of the Screening Visit to their health-care provider) of difficulty sleeping or daytime sleepiness while not experiencing SAR symptoms, and continue with these complaints
* Snoring associated with an enlarged uvula or other upper airway pathology
* Had episodes of snoring associated with gasping or choking
* Awakened suddenly, on more than 1 occasion during the month preceding the Screening Visit, with a gasping or choking feeling
* Requires the use of oral appliances at night for bruxism (teeth gnashing) or temporomandibular joint problems
* Diagnosis of asthma with daytime and nighttime asthma symptoms not controlled by short-acting beta-2 adrenoceptor agonists
* Dependence on nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* Currently undergoing a progressive course of immunotherapy (hyposensitization). Subjects on a regular maintenance schedule prior to the Screening Visit and who wish to remain on this schedule during the study are eligible for study inclusion; however, they may not receive hyposensitization treatment within 24 hours prior to any study visit
* Smokers or ex-smokers who have smoked within the previous 6 months
* Concomitant medical problem that may interfere with participation in the study, eg, repeated migraine episodes, uncontrolled convulsive disorders.
* Any of the following clinical conditions: Active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, systemic viral infections or ocular herpes simplex.
* Subjects participating in any other clinical study(ies).
* Subjects allergic to or with a sensitivity to the study drug or its excipients.
* Subjects who are night-shift workers or do not have a standard "asleep at night/awake during the day" cycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray: Mometasone Furoate Nasal Spray; 50 mcg/spray: self-administered, two sprays per nostril (ie, 200 mcg), once daily (each morning), for 28 days.
- Placebo Nasal Spray.: Matching placebo nasal spray. Two sprays per nostril once daily, for 28 days.
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray.
Started | 267 | 134
Completed | 254 | 131
Not Completed | 13 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-compliance with protocol | 6 | 1
Not completed — Administrative | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray. | Total
Number analyzed (Participants) | 267 | 134 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 259 | 132 | 391
  >=65 years | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (12.8) | 35.1 (11.8) | 35.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 85 | 255
  Male | 97 | 49 | 146

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of the AM-PRIOR-reflective (Participant's Status Over the Previous 12 Hours) Total Nasal Symptoms Severity Score (TNSS) Averaged Over the Last 7 Days of Treatment From the Baseline Score.
Description: The TNSS score included the sum of nasal congestion/stuffiness, rhinorrhea/nasal discharge, sneezing, and nasal itching, each scored on a scale of 0 = absent, 1 = mild, 2 = moderate, 3 = severe. The TNSS score could range from 0 to 12.
  NOTE: Least square means and standard errors were obtained from an ANCOVA model with the treatment effect and the variable specific Baseline as a covariate.
Time Frame: Average of the last 7 days of treatment
Population: Modified Intent-to-Treat (MITT) Population: all randomized subjects with any post-baseline data and without concomitant medications that could significantly bias the co-primary endpoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray.
Number analyzed (Participants) | 248 | 131
Units on a scale
  Change from Baseline in TNSS score | -3.77 (0.19) | -3.07 (0.26)
  Baseline TNSS score | 9.10 (0.10) | 9.12 (0.14)

2. Primary Outcome: Mean Change From Baseline (Day 1/Visit 3) in the Sleep Problems Index II (SLP9) Score From the Medical Outcome Study Sleep Scale (MOS-SS) at the Day 29 Visit.
Description: Following Visit 2 (Screening), at Baseline, Day 15, and Day 29 visits, participants needed to complete the MOS-SS questionnaire with scores from 1 = all of the time to 6 = none of the time, according to their frequency of occurrence during the previous week. The analysis endpoint MOS-SS Sleep Problems Index II (SLP9) score was derived from MOS-SS questionnaire and scaled from 0 = none of the time to 100 = all of the time.
  NOTE: Least squares means and standard errors were obtained from an ANCOVA model with the treatment effect and the variable specific Baseline as a covariate.
Time Frame: 29 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray.
Number analyzed (Participants) | 243 | 126
Units on a scale
  Change from baseline in SLP9 score | -26.1 (1.38) | -25.8 (1.90)
  Baseline SLP9 Score | 68.6 (0.86) | 69.2 (1.20)

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray.
Serious Adverse Events (participants affected / at risk) | 1/267 | 0/134
Other Adverse Events (participants affected / at risk) | 10/267 | 7/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=267) | Placebo Nasal Spray. (N=134)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=267) | Placebo Nasal Spray. (N=134)
Headache (Nervous system disorders) | 10 (16) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is not allowed to release any interim results of the Study without prior consent of the sponsor, and must provide 45 days written notice to the sponsor prior to public release to permit the sponsor's review. The PI can use the study results for his/her own teaching, research, and publication purposes only, not for commercial purposes, except as authorized by the sponsor. No publication shall contain any trade secret or proprietary/confidential information of the sponsor.